CLINICAL TRIAL: NCT06979076
Title: A Phase Ib Study of the Selective PKC-β Inhibitor MS-553 in Patients With Refractory or Relapsed Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: A Phase Ib Study of the Selective PKC-β Inhibitor MS-553 in Patients With Refractory or Relapsed CLL/SLL
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MingSight Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS-553-201-CLL
Record Dates: First submitted 2025-05-02; First posted 2025-05-18 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: CLL (Chronic Lymphocytic Leukemia); SLL (Small Lymphocytic Lymphoma)
MeSH Terms: conditions — Leukemia, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MS-553, dose schedule 1 (DS1) (Experimental)
  Interventions: Drug: MS-553, DS1
- MS-553, dose schedule 2 (DS2) (Experimental)
  Interventions: Drug: MS-553, DS2

INTERVENTIONS:
Drug: MS-553, DS1 — Oral, Dose Schedule 1
  Arms: MS-553, dose schedule 1 (DS1)
Drug: MS-553, DS2 — Oral, Dose Schedule 2
  Arms: MS-553, dose schedule 2 (DS2)

SUMMARY:
A Phase Ib Study of the Selective PKC-β Inhibitor MS-553 in Patients with Refractory or Relapsed Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Diagnosis of CLL or SLL:

   1. History of histologically documented CLL or SLL that meets iwCLL diagnostic criteria according to the 2018 guidelines, and
   2. Indication for treatment as defined by the 2018 iwCLL guidelines, or the need for disease reduction prior to allogeneic transplantation.-

Exclusion Criteria:

1. Current transformation of CLL/SLL non-Hodgkin lymphoma or Hodgkin lymphoma.
2. Active and uncontrolled autoimmune cytopenia(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The occurrence of AEs and SAEs, with abnormal laboratory tests results, abnormal physical examination findings, abnormal vital signs, and abnormal ECG readings | Through study completion, an average of 2 years